CLINICAL TRIAL: NCT04129216
Title: The Effects of Short-term Preoperative Treatment With Hormonal Therapy on Gene Profiles in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Agendia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00130428
Record Dates: First submitted 2019-05-17; First posted 2019-10-16 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; genomic assay; hormone therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Letrozole; exemestane

STUDY DESIGN:
Intervention Model Description: Patients will start the hormone therapy before surgery; the investigators look for the genomic profiles of the tumor before and after chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Tamoxifen arm (Experimental): for premenopausal patients
  Interventions: Drug: Tamoxifen Citrate; Diagnostic Test: Blueprint; Diagnostic Test: Mammaprint
- Letrozole arm (Experimental): for postmenopausal patients
  Interventions: Drug: Letrozole; Diagnostic Test: Blueprint; Diagnostic Test: Mammaprint
- Exemestane arm (Experimental): for postmenopausal patients
  Interventions: Drug: Exemestane; Diagnostic Test: Blueprint; Diagnostic Test: Mammaprint

INTERVENTIONS:
Drug: Tamoxifen Citrate — 10mg administered daily. Patients take this drug for 2-6 weeks
  Other Names: Soltamox
  Arms: Tamoxifen arm
Drug: Letrozole — 2.5mg is administered daily. Patients take this drug for 2-6 weeks
  Other Names: Femara
  Arms: Letrozole arm
Drug: Exemestane — 25mg is administered daily. Patients take this drug for 2-6 weeks.
  Other Names: Aromasin
  Arms: Exemestane arm
Diagnostic Test: Blueprint — studies the genomics of the tumor and tumor behavior
Diagnostic Test: Mammaprint — studies the genomics of the tumor

SUMMARY:
The investigators would like to study the genetic and molecular outcomes that results after a short term neoadjuvant hormonal therapy on patients with breast cancer.

DETAILED DESCRIPTION:
Breast cancer is among the most common malignancies in women in the United States. Over the years breast cancer management have dramatically developed from the extensive surgical approach toward the breast conservative approach. This was mainly due to the introduction of chemotherapy and hormonal therapy. Hormonal therapy in particular has been shown to improve the oncological outcomes of the breast cancer. However, while this is well documented in the clinical outcomes. Little is known in regards what happens on the genetic level. As such in this study the investigators would like to study the genetic and molecular outcomes that results after a short term neoadjuvant hormonal therapy on patients with breast cancer.

The hypothesis of this study is that short-term, preoperative hormonal treatment will induce genetic changes associated with reduced proliferation, including lower Ki67 expression, and changes in Estrogen Receptor (ER) and Progesterone Receptor (PR) expression. The data from such investigation will be very helpful in advancing the individualized care to women with breast cancer.

ELIGIBILITY:
Inclusion criteria

* Treatment-naïve, histologically confirmed invasive ductal breast cancer between stages 1 to 3.
* Co-enrollment in the FLEX Registry
* Estrogen Receptor Positive (ER+) Progesterone Receptor Positive (PR+) confirmed hormone receptor status measured by immunohistochemistry (IHC)
* Patients should understand patients' condition and be able to give informed consent to participate

Exclusion criteria

* History of hormonal therapy, chemotherapy, radiation therapy, or novel therapy to treat the current breast cancer.
* Allergic reactions/hypersensitivity to tamoxifen, letrozole, or exemestane or any of the ingredients of these drugs.
* Any contraindication to hormonal therapy, such as history of thromboembolic disease or uterine cancer.
* Patients without invasive disease (stage 0)
* Patients with metastatic breast cancer(stageIV)
* Patients that are Human Epidermal Growth Factor 2+(HER2+) by IHC/Fluorescence in situ hybridization (FISH).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Habibi, MD, Principal Investigator — Johns Hopkins Bayview
Locations (1):
- Johns Hopkins Bayview Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suman VJ, Ellis MJ, Ma CX. The ALTERNATE trial: assessing a biomarker driven strategy for the treatment of post-menopausal women with ER+/Her2- invasive breast cancer. Chin Clin Oncol. 2015 Sep;4(3):34. doi: 10.3978/j.issn.2304-3865.2015.09.01. PMID 26408301

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamoxifen Arm | Letrozole Arm | Exemestane Arm
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen Arm | Letrozole Arm | Exemestane Arm | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Customized [Number; unit: participants]
  below 55 | 7 | 0 | 0 | 7
  55 and above | 3 | 10 | 10 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 29
  Male | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 6 | 5 | 4 | 15
  African American | 4 | 5 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Expression of Ki67 Measured by Immunohistochemistry (IHC)
Description: This is a measure of tumor proliferation, and will be determined at baseline and at time of surgery.
Time Frame: Baseline and at Time of surgery up to 6 weeks after the start of hormone therapy
Measure: Mean (Standard Deviation); unit: Change in percentage expression of ki 67
Arm/Group | Tamoxifen Arm | Letrozole Arm | Exemestane Arm
Number analyzed (Participants) | 10 | 10 | 10
Change in percentage expression of ki 67 | -3.6 (1.06) | -5.1 (1.82) | -4.2 (1.71)

2. Secondary Outcome: Number of Participants With Low or High Score in MammaPrint
Description: Mammaprint risk score is binary (high risk of recurrence or low risk of recurrence).
Time Frame: Baseline and at Time of surgery (up to 6 weeks)
Measure: Count of Participants; unit: Participants
Groups:
- Tamoxifen Arm: for premenopausal patients Tamoxifen Citrate: 10mg administered daily. Patients take this drug for 2-6 weeks Blueprint: studies the genomics of the tumor and tumor behavior Mammaprint: studies the genomics of the tumor
- Letrozole Arm: for postmenopausal patients Letrozole: 2.5mg is administered daily. Patients take this drug for 2-6 weeks Blueprint: studies the genomics of the tumor and tumor behavior Mammaprint: studies the genomics of the tumor
- Exemestane Arm: for postmenopausal patients Exemestane: 25mg is administered daily. Patients take this drug for 2-6 weeks. Blueprint: studies the genomics of the tumor and tumor behavior Mammaprint: studies the genomics of the tumor
Arm/Group | Tamoxifen Arm | Letrozole Arm | Exemestane Arm
Number analyzed (Participants) | 10 | 10 | 10
Participants
  low risk mammaprint score at baseline | 5 | 7 | 5
  high risk mammaprint score at baseline | 5 | 3 | 5
  low risk mammaprint score at time of surgery (up to 6 weeks) | 7 | 8 | 7
  high risk mammaprint score at time of surgery (up to 6 weeks) | 3 | 2 | 3

3. Secondary Outcome: Median Percent of Tissue ER Positive
Description: Median percent of tissue ER positive in matched tissue measured by Immunohistochemistry (IHC)
Time Frame: Baseline and at Time of surgery (up to 6 weeks)
Measure: Median (Full Range); unit: percent of tissue ER positive
Arm/Group | Tamoxifen Arm | Letrozole Arm | Exemestane Arm
Number analyzed (Participants) | 10 | 10 | 10
percent of tissue ER positive
  Baseline median percent of tissue ER positive | 98 [67 to 100] | 93 [76 to 99] | 95 [50 to 100]
  Time of surgery (up to 6 weeks) median percent of tissue ER positive | 95 [90 to 95] | 95 [60 to 97] | 95 [50 to 100]

4. Secondary Outcome: Median Percent of Tissue PR Positive
Description: Median percent of tissue PR positive in matched tissue measured by Immunohistochemistry (IHC)
Time Frame: Baseline and at Time of surgery (up to 6 weeks)
Measure: Median (Full Range); unit: percent of tissue PR positive
Arm/Group | Tamoxifen Arm | Letrozole Arm | Exemestane Arm
Number analyzed (Participants) | 10 | 10 | 10
percent of tissue PR positive
  Baseline median percent of tissue PR positive | 97 [67 to 100] | 33 [0 to 95] | 83 [0 to 100]
  Time of surgery (up to 6 weeks) median percent of tissue PR positive | 90 [75 to 95] | 0 [0 to 71] | 7 [0 to 35]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Description: all adverse effects were collected
Arm/Group | Tamoxifen Arm | Letrozole Arm | Exemestane Arm
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
small number of participants

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-18): https://cdn.clinicaltrials.gov/large-docs/16/NCT04129216/Prot_SAP_000.pdf